CLINICAL TRIAL: NCT01690936
Title: Effects of Chronic Almond Consumption at Meals or as Snacks on Appetite, Intake, Body Weight, Glycemia, Insulinemia and Lipids in Healthy Adults.
Brief Title: Metabolic Effects of Almond in the Longer-term Study
Acronym: MEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Prof Foods and Nutrition, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 055-022; Snacking study (Other Grant/Funding Number: Almond Board of California)
Record Dates: First submitted 2012-09-12; First posted 2012-09-24 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Obesity
Keywords: Almonds; Body weight; Snacking
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Breakfast (Experimental): Almonds (43g/day) were consumed with breakfast for four weeks.
  Interventions: Dietary Supplement: Almonds 43g/day
- Morning snack (Experimental): Almonds (43g/day) were consumed alone as morning snacks for four weeks.
  Interventions: Dietary Supplement: Almonds 43g/day
- Lunch (Experimental): Almonds (43g/day) were consumed with lunch for four weeks.
  Interventions: Dietary Supplement: Almonds 43g/day
- Afternoon snack (Experimental): Almonds (43g/day) were consumed alone as afternoon snacks for four weeks.
  Interventions: Dietary Supplement: Almonds 43g/day
- Control no nuts (No Intervention): Avoided all nuts and seeds

INTERVENTIONS:
Dietary Supplement: Almonds 43g/day — 43 grams of almonds were supplemented to the 4 intervention arms but eaten at different times of day (with meals or alone as snacks) for 4 weeks. Control group was asked to avoid all nuts/seeds during the study period
  Arms: Afternoon snack; Breakfast; Lunch; Morning snack

SUMMARY:
Identifying snacks that do not contribute to positive energy balance is crucial in weight management. The satiating effects of almonds, coupled with their convenience and palatability make them a promising weight management aid. Therefore, this study aimed to examine the effects of almond consumption with meals versus snacks on outcomes such as appetite, energy intake, body weight, as well as blood glucose, insulin and lipid responses.

DETAILED DESCRIPTION:
Experiment protocol and measurements

i) Oral glucose tolerance test (OGTT) sessions

At baseline, participants attended a session where a standard OGTT with drinks containing 75 grams dextrose was performed following an overnight fasting. Serum glucose and insulin concentrations were measured at 0 and 120 minutes of the session. During the same session, height, weight (Tanita), body fat (air displacement plethysmography, BOD POD), waist circumference, and blood pressure were measured. Participants also completed a 24-hour dietary recall using a multi-pass interview method and standard questionnaires that assessed personality, eating behavior and habitual physical activity levels during the OGTT session. After the completion of this session, participants were asked to record their hourly appetite sensations, measured as "hunger", "fullness" and "desire to eat" on visual analog scales, during waking hours for a day before attending the next (clinical) visit. Participants repeated this session after four weeks of almond consumption.

ii) Acute feeding sessions

Within a week following the OGTT session, participants returned for an acute-feeding session, after an overnight fasting of at least 10 hours. This session began between 7:00 am and 8:00 am, and lasted for approximately 515 minutes. Upon arrival, an indwelling arm catheter was placed in the upper arm for blood sample collection. Participants rested for 15 minutes after catheter placement, before a baseline blood sample was drawn. Immediately after the first blood sample collection, a standard breakfast was served, and participants were instructed to consume the entire portion within 10 minutes. Subsequent blood samplings were performed at 15, 45, 60, 90, 120, 180, and 240 minutes after the breakfast, before a standard lunch was provided to the participants. Again, participants were given 10 minutes to consume the lunch, before blood samples were taken at similar intervals again (at 265, 295, 310, 340, 370, 430, and 490 minutes of the session). Participants randomized into the BF and LN groups received 43 grams of almonds together with their meals, while the MS and AS groups consumed 43 grams of almonds 120 minutes after breakfast and lunch respectively. Participants also recorded their "hunger", "fullness", and "desire to eat" sensations when blood samples were taken. During the acute-feeding session, activities that may alter appetite sensations (e.g. sleeping and watching movies containing food cues) were prohibited. Postprandial glucose, insulin and triacylglycerol concentrations were measured for all 15 samples collected from each participant. Participants in all almond groups group were also asked to rate their likings for the almonds they ingested using a general label magnitude scale, and their action responses to almonds using the "food action rating scale", a visual analog scale ranging from "I would eat the almonds only if I were forced to" to "I would eat this food every opportunity I had" anchored to the 2 extremes. This session was repeated again after four weeks of almond supplementation.

iii) Weekly follow-ups

Following the baseline acute-feeding session, participants were asked to consume 43 grams of almonds every day at times based on their group randomization. The CL group was instructed to avoid all nuts and seeds in the diet during the study period. All almonds were dry-roasted and lightly salted, and were pre-weighed and per-packaged for convenience. Except for the permission to adjust dietary intake due to almond supplement, participants were asked to maintain their dietary intakes and physical activity levels. A ruse (breath analysis) was introduced in order to enhance the compliance of participants to consuming almonds at the designated times of day. Compliance to almond consumption was assessed through fasting plasma α-tocopherol. Participants attended weekly visit (week-1, 2 and 3) after an overnight fasting, during which body weight was recorded and compliance to study protocol reinforced. During the week-2 visit, participants were also asked to complete a 24-hour dietary intake assessment using the multi-pass interview method and appetite sensation ratings on VAS at every waking hour for a day. On week-4, participants returned for OGTT and acute-feeding sessions as described above. The study protocol was approved by the Purdue University Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

* Not taking any medication known to affect glycemia, lipid metabolism or appetite
* Regular breakfast consumers
* Eat at least 5 meals a day
* Weight stable
* Either one of the 6 conditions
* BMI 27-35
* Family history of diabetes
* Fasting glucose between 6.1-6.9 mmol/L
* 2-hour glucose 7.8-11.1 mmol/L
* blood pressure >130/85 mmHg
* Waist >102cm (men) and >88cm (women)

Exclusion Criteria:

* Nut allergy
* Not willing to eat test foods and almonds

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose, insulin and lipids | 490 minutes
  Responses of these parameters to a standard breakfast and a standard lunch for all participants, plus almonds at designated times according to group randomization.
Anthropometric measurements | 4 weeks
  Changes in body weight, BMI, fat mass, waist circumference over 4 weeks
Fasting blood biochemistries | 4 weeks
  Fasting glucose, insulin and lipids at baseline, week-1, 2, 3 and 4
Dietary intake | 4 weeks
  Dietary intakes were assessed at baseline, week-2, and week-4 of study

SECONDARY OUTCOMES:
Blood pressure | Baseline and week-4
  Blood pressure measurements at baseline and final week of study
Appetite ratings | Baseline, week-2, and week-4
Postprandial appetite sensations | 490 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States